CLINICAL TRIAL: NCT01528241
Title: A Multi-center, Open-label Study in Elderly Healthy Volunteers and Elderly Patients With Major Depressive Disorder to Characterize the Regional Distribution of [11C] ABP688 in Brain by Positron Emission Tomography (PET)
Brief Title: Characterize the Regional Distribution of [11C] ABP688 in Brain by Positron Emission Tomography (PET)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CABP688A2102
Record Dates: First submitted 2012-02-03; First posted 2012-02-07 (Estimated); Last update posted 2020-12-08 (Actual); Status verified 2012-02

CONDITIONS: Depression
Keywords: ABP688; Tracer; Depression
MeSH Terms: conditions — Depression | interventions — 3-(6-methylpyridin-2-ylethynyl)cyclohex-2-enone-O-methyloxime

ARMS (1):
- ABP688 (Experimental): Elderly MDD patients and demography matched healthy volunteer
  Interventions: Drug: ABP688

INTERVENTIONS:
Drug: ABP688 — Carbon 11 labeled ABP688 will be administered intravenously as a slow intravenous push.

SUMMARY:
This study is designed to characterize the regional distribution of [11C] ABP688 in brain by positron emission tomography (PET).

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects 55-80 (inclusive)
* Subjects in good health

At screening:

* oral body temperature between 35-37.5C
* systolic blood pressure: 90-140 mm Hg
* diastolic blood pressure: 50-90 mm Hg
* pulse rate: 40-90 bpm
* Female subjects of child bearing potential must have been using a double-barrier local contraception
* Postmenopausal women must have had no menstrual bleeding
* Subjects must have weighed at least 50 kg
* All subjects must provide informed consent
* All subjects must have been able to communicate well with investigator

Specific to Major depression disorder (MDD)

Patients had to show following level of symptomatology:

* HAM-D (17-item scale) > 16
* CGI > 4 (moderately ill)

Exclusion Criteria:

Specific criteria for healthy volunteers:

- Presence and/or history of clinically significant major neurological or psychiatric disorder

Specific criteria for MDD patients:

* Presence and/or history of a clinically significant major neurological or psychiatric disorder other than MDD or generalized anxiety disorder
* Axis I co-morbidity was excluded except anxiety spectrum disorders

Criteria for both:

* Smokers
* Pregnancy
* Subjects with history of or symptoms/complaints consistent with mild cognitive impairment
* Use of any psychotropic prescription drugs
* Coffee consumers more than 6 cups/day
* Participation in any clinical investigation
* Donation or loss of 400 mL or more of blood
* Significant illness within 2 weeks prior to dosing
* A known hypersensitivity to study drug
* MRI scan that showed evidence of stroke
* Any surgical or medical condition which might have significantly altered distribution
* Clinical evidence of any abnormal lab value
* History of immunodeficiency disease
* Positive Hepatitis B surface antigen
* Presence of contraindications to PET scan investigations- Presence of contraindications to MRI investigations
* Evidence from an Allen test of incomplete communication
* History of drug or alcohol abuse
* Current use of anticonvulsant
* Significant radiation exposure

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2008-08; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Binding of [11C] ABP688 to mGlu5 receptors | Day 1
  Binding of [11C]ABP688 will be determined using positron emission tomography (PET) for up to 90 minutes
Blood levels of [11C] ABP688 | Day 1, up to 60 minutes
  Blood samples (up to 19 time points via indwelling catheter) will be collected for the determination of [11C] ABP688. Specific times are recorded at the clinical site.

SECONDARY OUTCOMES:
Difference in [11C]ABP688 binding to mGlu5 receptors | Day 1
  Using data generated as described above, data will be analyzed to determine if there are difference in binding between healthy volunteers and patients.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (2):
- United States (2):
  - Novartis Investigative Site, New York, New York
  - Novartis Investigative Site, Pittsburgh, Pennsylvania

REFERENCES:
- See also: Results for CABP688A2102 can be found on the Novartis Clinical Trial Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=5125